CLINICAL TRIAL: NCT05180071
Title: A Post-market Study Evaluating Clinical and Radiographic Outcomes of Total Elbow Arthroplasty With TEMA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Limacorporate S.p.a (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-02
Record Dates: First submitted 2021-12-17; First posted 2022-01-06 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-09

CONDITIONS: Total Elbow Arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TEMA elbow arthroplasty (Experimental)
  Interventions: Device: TEMA elbow system

INTERVENTIONS:
Device: TEMA elbow system — Total elbow replacement

SUMMARY:
TEMA elbow system is a CE marked medical device, and within this clinical trial it is used according to its intended use. This is a Post Marketing Clinical Follow Up trial, with the main aim to collect evidences on the outcome data on this product, by analysing clinical scoring systems, radiographs and adverse event records within five years after the surgery, and thus to assess the short-term performance and safety of this implant.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's age ≥ 18 years old.
2. Patient has given written informed consent to participate to the trial and to his/her personal data processing
3. According to the device indications for use, patient suffers from disability due to one or more of the following:

   * Elbow joint destruction which significantly compromises the activities of daily living
   * Non-Inflammatory degenerative joint disease including osteoarthritis and avascular necrosis with hemophilia.
   * Rheumatoid arthritis or degenerative arthritis with incapacitating pain
   * Correction of severe functional deformity.
   * Treatment of acute or chronic fractures with distal humerus epicondyle involvement.
   * Post-traumatic lesions or bone loss contributing to elbow instability or loss of motion
   * Any other medical reason that the investigator determine that subject is a good candidate for a total elbow arthroplasty
4. Patient has undergone a total elbow arthroplasty, receiving TEMA prosthesis.
5. Patient is able to comply with the study protocol.

Exclusion Criteria:

A patient will be excluded from the study participation if he/she meets any of the following criteria:

1. Patient is affected by one or more of the conditions that are stated as TEMA contraindications for use, which are:

   * Local or systemic infection;
   * Septicemia;
   * Persistent acute or chronic osteomyelitis.
   * Uncooperative patient or patient with neurologic disorders who are incapable of following directions;
   * Osteoporosis;
   * Metabolic disorders which may impair bone formation;
   * Rapid joint destruction, marked bone loss or bone resorption.
2. Patient suffers from a diaphyseal fracture
3. For female patients, current pregnancy and/or lactation or planning a pregnancy.
4. Only for patients implanted with the unlinked configuration of TEMA prosthesis, the intraoperative testing showed a bad quality of medial and lateral elbow ligaments.
5. Patient is enrolled in another investigational drug/device study that in the opinion of the Investigator could interfere with this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Oxford Elbow Score improvement at three ears FU | 2 years Follow up
  Functional change in Oxford Elbow Score (OES) from preoperative (baseline) to 2 years of follow-up.

IPD SHARING:
Plan to Share IPD: No